CLINICAL TRIAL: NCT05471063
Title: Clinical Study of Amphotericin B Colloidal Dispersion (ABCD) in the Treatment of Cryptococcal Meningitis
Brief Title: Clinical Study of ABCD in the Treatment of Cryptococcal Meningitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Group Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, LI Taisheng, Director in department of Infectious Diseases, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-ABCD-K09
Record Dates: First submitted 2022-07-01; First posted 2022-07-22 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Cryptococcal Meningitis
Keywords: cryptococcal meningitis; Amphotericin B Colloidal Dispersion; non-HIV patients
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — Amphotericin B; Injections; Flucytosine; Fluconazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABCD treatment (Experimental): In this single-arm research, patients were treated with ABCD 3.0-4.0 mg/kg/d (subject to adjustment, maximum dose not exceeding 6.0 mg/kg/d) combined with flucytosine 100 mg/kg/d for induction therapy of cryptococcal meningitis. The course of induction therapy is at least four weeks. Then, patients were treated with Fluconazole (400-600 mg/d) ± flucytosine (100 mg/kg/d) for consolidation therapy for at least 6 weeks.
  Interventions: Drug: Amphotericin B Colloidal Dispersion; Drug: flucytosine; Drug: fluconazole

INTERVENTIONS:
Drug: Amphotericin B Colloidal Dispersion — Amphotericin B Colloidal Dispersion 3.0-4.0 mg/kg/d (subject to adjustment, maximum dose not exceeding 6.0 mg/kg/d) . The course of induction therapy is at least four weeks.
  Other Names: Amphotericin B Cholesteryl Sulfate Complex for Injection
Drug: flucytosine — Flucytosine 100 mg/kg/d for induction therapy and consolidation therapy of cryptococcal meningitis. The course of induction therapy is at least four weeks, and consolidation therapy for at least 6 weeks.
  Other Names: fluorocytosine
Drug: fluconazole — Fluconazole (400-600 mg/d) for consolidation therapy for at least 6 weeks.
  Other Names: Diflucan

SUMMARY:
To evaluate the efficacy and safety of ABCD in the treatment of cryptococcal meningitis in non-HIV patients at week 4, the end of induction therapy, week 10 and the end of consolidation therapy.

DETAILED DESCRIPTION:
This study is a multi-center, single-arm clinical study. The objective is to evaluate the efficacy and safety of ABCD in the treatment of cryptococcal meningitis in non-HIV patients. Qualified subjects shall receive cryptococcus induction therapy with ABCD combined with flucytosine for at least 4 weeks, or termination of treatment early at the investigator's discretion. Efficacy and safety are followed up at week 4 (day 28), the end of induction therapy, week 10 (day 70) and the end of consolidation therapy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old and ≤70 years old, no gender limitation;
* Diagnosis of cryptococcal meningitis (with or without other cryptococcal lesions) based on CSF culture and/or CSF ink staining smear and/or CSF antigen testing;
* The researcher believes that patients can benefit from participating in this study;
* The subjects voluntarily participated in the study and signed the informed consent.

Exclusion Criteria:

* Patients with other invasive fungal diseases;
* HIV infected patients;
* Patients who received intravenous polyene treatment within the past 6 months;
* Allergic to Amphotericin B Colloidal Dispersion or other ingredients in this product;
* Patients with abnormal liver function [aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >＝5 times the upper limit of normal value (ULN) without total bilirubin elevation, or ALT or AST >＝ 3 times ULN with total bilirubin >＝ 1.5 times];
* Patients with impaired renal function (renal function index blood creatinine (Cr) is more than 2 times higher than ULN, or 24-hour urine creatinine clearance rate （Ccr） is less than 50ml/min), or patients requiring/undergoing hemodialysis or peritoneal dialysis;
* Pregnant women, breast-feeding women and women of childbearing age who were unable to take effective contraceptive measures during the study period;
* Conditions considered unsuitable for the study by the investigator, such as concomitancy of severe organ insufficiency, clinically significant laboratory abnormalities, comprehension or compliance problems, etc.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-22 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with complete or partial response at the end of induction therapy | From enrollment to the end of induction therapy (about 4-6 weeks)
  Complete response: live during the observation period, patients with cryptococcus meningitis all the clinical signs and symptoms disappeared, a significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
  Partial response: patient survival during the observation period, cryptococcal meningitis clinical signs and symptoms improved, all the significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.

SECONDARY OUTCOMES:
Proportion of patients with complete or partial response at 4 weeks | At the 4 weeks of treatment
  Complete response: live during the observation period, patients with cryptococcus meningitis all the clinical signs and symptoms disappeared, a significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
  Partial response: patient survival during the observation period, cryptococcal meningitis clinical signs and symptoms improved, all the significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
Proportion of patients with complete or partial response at 10 weeks | At the 10 weeks of treatment
  Complete response: live during the observation period, patients with cryptococcus meningitis all the clinical signs and symptoms disappeared, a significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
  Partial response: patient survival during the observation period, cryptococcal meningitis clinical signs and symptoms improved, all the significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
Proportion of patients with complete or partial response at the end of consolidation therapy | At the end of the consolidation therapy (about 12 weeks)
  Complete response: live during the observation period, patients with cryptococcus meningitis all the clinical signs and symptoms disappeared, a significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
  Partial response: patient survival during the observation period, cryptococcal meningitis clinical signs and symptoms improved, all the significant reduction in the cerebrospinal fluid cryptococcal antigen test results and/or CSF cryptococcus training and/or ink staining (two consecutive tests, one week interval) results overcast, and abnormal head MRI/CT (if exist in baseline) improved or stable.
Cryptococcus antigen titer | 1,2,3,4,10 weeks
  Diachronic changes in antigenic titers of Cryptococcus
Duration of the cryptococcal meningitis | At the end of the consolidation therapy (about 12 weeks)
  The time from this hospitalization to the end of consolidation therapy.
Adverse events | about 12 weeks
  Incidence and severity of adverse events during treatment, evaluated according to NCI-CTCAE Ver. 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Taisheng Li, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No